CLINICAL TRIAL: NCT03920644
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 3 Study of the Safety and Efficacy of Defender Pharmaceuticals Inc, (DPI)-386 Nasal Gel on Ocean-Going Vessels for the Prevention and Treatment of Nausea Associated With Motion Sickness
Brief Title: Study of the Safety and Efficacy of DPI-386 Nasal Gel on Ocean-Going Vessels
Acronym: INSCOP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Naval Aeromedical Research Unit, Dayton (U.S. Federal Agency)
Responsible Party: Principal Investigator, Matthew Doubrava, Senior Medical Officer, Aeromedical department Head, Naval Aeromedical Research Unit, Dayton
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NAMRUD.2018.0002 Field Trial
Record Dates: First submitted 2019-04-03; First posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Prevention of Nausea Associated With Motion Sickness; Treatment of Nausea Associated With Motion Sickness
Keywords: Motion Sickness, INSCOP, Scopolamine, Defender, NAMRU
MeSH Terms: conditions — Motion Sickness | interventions — Scopolamine; tyramine-deoxysorbitol; Transdermal Patch

STUDY DESIGN:
Intervention Model Description: The study will include 120 subjects per arm, for a total of 360 subjects (n=360). A double-dummy design will be used to mask the treatment assignment. All subjects will receive both a patch and nasal gel: DPI-386 Nasal Gel + placebo patch, placebo nasal gel + placebo patch, or TDS patch + placebo nasal gel.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DPI-386 Nasal Gel (Experimental): Receives Active Nasal Gel 2 times per treatment day
  Interventions: Drug: Scopolamine; Drug: Placebo Patch
- Placebo nasal gel (Placebo Comparator): Receives Nasal Gel 2 times per treatment day
  Interventions: Drug: Placebo Patch; Drug: Placebo Gel
- TDS Patch (Active Comparator): Receives one patch per treatment.
  Interventions: Drug: Scopolamine Transdermal Patch [Transderm Scop]; Drug: Placebo Gel

INTERVENTIONS:
Drug: Scopolamine Transdermal Patch [Transderm Scop] — Current Motion Sickness treatment, 1 patch behind the ear.
  Other Names: TDS, Patch
  Arms: TDS Patch
Drug: Scopolamine — IND, up to 6 administration of intranasal gel.
  Other Names: DPI-386
  Arms: DPI-386 Nasal Gel
Drug: Placebo Patch — Placebo Patch, 1 patch behind the ear.
  Arms: DPI-386 Nasal Gel; Placebo nasal gel
Drug: Placebo Gel — Placebo Gel,up to 6 administration of intranasal gel.
  Arms: Placebo nasal gel; TDS Patch

SUMMARY:
This multi-site Phase 3 clinical trial is a randomized, double-blind, placebo-controlled study to identify the safety and efficacy of DPI 386 nasal gel (intranasal scopolamine gel) for the prevention and treatment of nausea associated with motion sickness. The study will be conducted aboard military ships undergoing military operations or aboard commercial boats rented for the study to obtain data in a real world environment. The study will have three arms: DPI-386 nasal gel, placebo nasal gel, and Transderm Scop® (1.0 mg/72 hours; transdermal scopolamine patch [TDS], the current standard of care for the treatment of motion sickness). The study will include 120 subjects per arm, for a total of 360 subjects (n=360). A double-dummy design will be used to mask the treatment assignment. All subjects will receive both a patch and nasal gel: DPI-386 Nasal Gel + placebo patch, placebo nasal gel + placebo patch, or TDS patch + placebo nasal gel.

ELIGIBILITY:
Inclusion Criteria:

* 1. Provision of signed and dated Informed consent document (ICD). 2. Stated willingness to comply with all study procedures and availability for the duration of the study.

  3. Male or female, aged 18 to 59 (inclusive). 4. Tricare health insurance beneficiary. All potential subjects must be able to provide a current military Identification (ID) or Department of Defense (DOD) dependent ID to be viewed by the research staff prior to signing the ICD.

  5. At least minimally susceptible to provocative motion as evidenced by a minimum score of 3.0 on the MSSQ.

  6. In good general health as evidenced by medical history with no recent history or current diagnosis of clinical problems as assessed by the research staff.

  7. Ability to take intranasal medication and willingness to adhere to the study schedule and time constraints.

  8. For females of child-bearing potential: willingness to provide a urine sample for the hCG pregnancy test during the Screening Visit and each day of the Treatment Period. Test must be negative or the subject will be excluded from the study. Note: Women of non-childbearing potential are defined as those who are non-surgically sterile (i.e., without menses for at least 12 consecutive months) or surgically sterile (i.e., those who underwent a hysterectomy with or without oophorectomy, fallopian tube ligation, and endometrial ablation).

  9. Agreement to adhere to the following lifestyle compliance considerations:
  1. Refrain from consumption of grapefruit and any substance containing grapefruit for seven days prior to, during, and for seven days after the Treatment Period.
  2. Abstain from alcohol for 24 hours prior to first dose of study medication and during the Treatment Period.
  3. Note: there will be no restriction on caffeine or nicotine use during the study; however, the actual use of these substances will be recorded as part of the CEBQ.

     Exclusion Criteria:
* 1. Pregnancy, lactation, or positive urine pregnancy test at any time. 2. Known allergic reactions to any drugs. 3. Currently prescribed any of the following medication types: any form of scopolamine (including Transderm Scop®) within 5 days, belladonna alkaloids within 2 weeks, antihistamines (including meclizine) within 2 weeks, tricyclic antidepressants within 2 weeks (depending on reason taken), muscle relaxants and nasal decongestant within 4 days of Module 1.

  4. Hospitalization or significant medical event (to include childbirth) within the past six months.

  5. Treatment with another investigational drug or other intervention within the past 30 days.

  6. Having donated blood or plasma or suffered significant blood loss within the past 30 days.

  7. Having any of the following medical conditions within the last two years or if any of the following medical conditions were experienced more than two years ago and are deemed clinically significant by the PI or Study Physician:
  1. Any known drug allergies and/or severe year-round environmental allergies.
  2. Significant gastrointestinal disorder, asthma, or seizure disorders.
  3. History of vestibular disorders.
  4. History of narrow-angle glaucoma.
  5. History of urinary retention problems.
  6. History of alcohol or drug abuse.
  7. Nasal, nasal sinus, or nasal mucosa surgery.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 320 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Determine the efficacy of DPI-386 nasal gel compared to the TDS patch and placebo nasal gel in the prevention and treatment of nausea associated with motion sickness. | Through study completion, an average of 1 year
  The efficacy endpoint will be determined by comparing the Motion Sickness Assessment Questionnaire (MSAQ)(scale 1-10) scores over the treatment period across all three treatment arms
Determine the safety of DPI-386 Nasal Gel compared to the TDS patch and placebo nasal gel with an emphasis on cognitive effects. | Through study completion, an average of 1 year
  the safety endpoint is the incidence of adverse events.

SECONDARY OUTCOMES:
Determine the efficacy of DPI-386 Nasal Gel compared to the TDS patch and the placebo nasal gel in severity of nausea. | Through study completion, an average of 1 year
  Severity of nausea will measured by the Nausea Assessment (VAS)(scale 1-9) over the treatment period.
Determine the safety of DPI-386 Nasal Gel as compared to the TDS patch and placebo nasal gel in terms of cognition. | Through study completion, an average of 1 year
  Safety in terms of cognition will be measured by Computer task.

CONTACTS AND LOCATIONS:
Locations (1):
- NAMRU Dayton, Dayton, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided